CLINICAL TRIAL: NCT06868784
Title: Investigation of the Relationship Between Executive Functions and Occupational Performance of Children With Duchenne Muscular Dystrophy
Status: Enrolling by invitation | Type: Observational
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Başak Çağla Arslan, Lecturer, Lokman Hekim University
Other Study IDs: 2023025
Record Dates: First submitted 2024-05-10; First posted 2025-03-11 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Executive Dysfunction; Occupational Problems; Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Duchenne muscular dystrophy
  Interventions: Other: Evaluations
- Healthy control group of children
  Interventions: Other: Evaluations

INTERVENTIONS:
Other: Evaluations — Evaluations of executive functions and occupational performance

SUMMARY:
The effects of Duchenne muscular dystrophy and its treatments on executive functions and occupational performance are under-mentioned in the literature. The researches believe that developmental and cognitive research is needed to identify interventions for children with DMD to identify and adapt to both individual and social environments, including self-care, productivity and leisure activities. Therefore, the aim of this study was to examine executive functions and occupational performance in children with DMD and compare them with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with DMD
* Volunteering to participate in the study by their parents and reading and signing the informed consent form

Exclusion Criteria:

* Having a neuromuscular disease other than DMD and/or another diagnosed neuromuscular disease accompanying DMD
* The family and/or the child has problems with cooperation in completing the assessments for any reason
* Difficulty understanding and speaking the Turkish language

Ages: 6 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All boys diagnosed with DMD between the ages of 6-12 years constitute the population of this study.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographic information form | one-time evaluation
Brooke upper extremity functional scale | one-time evaluation
  It will be used to assess the functional level of the upper limbs of children with DMD. The classification consists of six stages and progression from the first to the sixth stage indicates a decrease in the functionality of the upper limb.
Vignos lower extremity functional scale | one-time evaluation
  It will be used to assess the functional level of the lower limbs of children with DMD. The classification consists of ten stages and progression from the first to the tenth stage indicates a decrease in the functionality of the upper limb.
The Childhood Executive Functioning Inventory | one-time evaluation
  This 26-item scale consists of 4 subscales: working memory (9 items), planning (6 items), inhibition (6 items) and regulation (5 items). Working memory and planning sub-dimensions constitute the total score of "working memory" and inhibition and regulation sub-dimensions constitute the total score of "inhibition". As the score obtained from the scale increases, the child's executive functions weaken.
Canadian Occupational Performance Measure | one-time evaluation
  It will be used to assess children's occupational performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Patient data in this study will not be shared with other researchers. The results of the study will be shared after anonymizing the demographic information of DMD and healthy children.